CLINICAL TRIAL: NCT00979303
Title: The Adjunct Use of Non-Fluoroscopic Imaging Devices to Decrease Radiation Exposure During Ablation of Supraventricular Tachycardia
Brief Title: Using Non-Fluoroscopic Imaging Devices to Decrease Radiation Exposure During Ablation of Supraventricular Tachycardia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Christina Yumi Miyake, Fellow, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08110505
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: Supraventricular Tachycardia
Keywords: Pediatric; Electrophysiology; Ablation; Radiation; Devices; SVT
MeSH Terms: conditions — Tachycardia, Supraventricular

STUDY DESIGN:
Intervention Model Description: Intent to treat use of non fluoroscopic mapping system with traditional fluoroscopic mapping system during elective catheter ablation in children 8-17 with normal cardiac anatomy
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Control Patients - Undergo ablation procedures with radiation/fluoroscopy only
- Study Group (Experimental): Study Group Patients - Undergo ablation procedures using intracardiac echocardiography and 3D navigational system in addition to radiation.
  Interventions: Device: Intracardiac echocardiography and 3D navigational system

INTERVENTIONS:
Device: Intracardiac echocardiography and 3D navigational system — Patients assigned to the intervention group will receive both intracardiac echocardiography as well as a 3D navigational system in addition to fluoroscopy during their ablation procedure.
  Other Names: AcuNav Intracardiac Echocardiography; NavX 3D navigational system; CARTO 3D navigational system
  Arms: Study Group

SUMMARY:
The purpose of this study is to determine whether the additional use of non-fluoroscopic imaging modalities can decrease the use of radiation exposure during standard ablation procedures for supraventricular tachycardia (SVT) in children.

DETAILED DESCRIPTION:
The standard of care for children undergoing SVT ablation is radiation (fluoroscopy) to see the heart. Non fluoroscopic imaging tools have been utilized for adult atrial fibrillation procedures. These tools utilize magnetic fields to visualize the heart without using radiation. The purpose of this study was to determine if these 3D mapping tools could reduce radiation exposure during SVT ablation procedures could be performed using these 3D tools.

ELIGIBILITY:
Inclusion Criteria:

* Age >/=8
* Weight >/=25kg
* Structurally normal heart (no major cardiac defects)
* History of SVT
* No prior history of cardiac surgery or ablation

Exclusion Criteria:

* Congenital Heart Disease
* Prior history of cardiac surgery or ablation

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2009-01-09 (Actual); Primary Completion 2009-09-28 (Actual); Study Completion 2010-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Y. Miyake, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Result] Miyake CY, Mah DY, Atallah J, Oikle HP, Melgar ML, Alexander ME, Berul CI, Cecchin F, Walsh EP, Triedman JK. Nonfluoroscopic imaging systems reduce radiation exposure in children undergoing ablation of supraventricular tachycardia. Heart Rhythm. 2011 Apr;8(4):519-25. doi: 10.1016/j.hrthm.2010.12.022. Epub 2010 Dec 15. PMID 21167315
- Available data/document: Archived consent, protocol and analytic plan. — http://www.childrenshospital.org/ — Study completed prior to change in common rule. Requests should be directed to the investigation team at Boston Children's Hospital through mark.alexander@cardio.chboston.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Study Group
Started | 37 | 37
Completed | 37 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Study Group | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37 | 35 | 72
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 14.2 [8.0 to 20.5] | 14.7 [8.6 to 22.3] | 14.5 [8.0 to 22.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 17 | 19 | 36
Region of Enrollment [Number; unit: participants]
  United States | 37 | 37 | 74
Weight [Mean (Full Range); unit: kg] | 57.9 [27.4 to 92.2] | 59.1 [26.8 to 104.0] | 58.5 [26.8 to 104.0]
Height [Mean (Full Range); unit: cm] | 162 [126 to 190] | 162.2 [134 to 184] | 162.1 [126 to 190]
Chest circumference [Mean (Full Range); unit: cm] | 17.4 [12.5 to 24.5] | 17.5 [12 to 27] | 17.4 [12 to 27]
BSA [Mean (Full Range); unit: m^2] | 1.6 [1.0 to 2.2] | 1.6 [1.0 to 2.2] | 1.6 [1.0 to 2.2]
BMI [Mean (Full Range); unit: kg/m^2] | 21.4 [15.0 to 31.3] | 22.3 [14.9 to 41.7] | 21.9 [14.9 to 41.7]

OUTCOME MEASURES:

1. Primary Outcome: Total Fluoroscopy Time
Description: Total fluoroscopy time in minutes
Time Frame: During the Ablation procedure
Measure: Median (Full Range); unit: minutes
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 37 | 37
minutes | 18.3 [5.4 to 74.4] | 7.5 [0 to 52.9]

2. Secondary Outcome: Total Radiation Exposure
Description: Total radiation exposure measured in mGy
Time Frame: During Ablation Procedure
Measure: Median (Full Range); unit: mGy
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 37 | 37
mGy | 387 [68 to 2701] | 110 [0 to 3026]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were evaluated in all patients during the study, prior to discharge and in follow up at 1 month and 1 year after the procedure.
Arm/Group | Control Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 8/37 | 6/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=37) | Study Group (N=37)
Hematoma (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3) — Groin hematoma
bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Brochospasm after adenosine
Headache (Nervous system disorders) | 1 (1) | 1 (1) — Headache
Vasovagal syncope (Nervous system disorders) | 0 (0) | 1 (1) — Vasovagal syncope
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) — Neuropathy
Mechanical trauma to pathway (Cardiac disorders) | 0 (0) | 1 (1) — Trauma to pathway
Groin Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Groin pain 1 week after discharge
Skin abrasion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Skin abrasion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes